CLINICAL TRIAL: NCT00940056
Title: Totally Endoscopic Ablation of Atrial Fibrillation
Acronym: TEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Anders Ahlsson, MD PHD, Region Örebro County
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UHOrebro; NCT01047228 (obsolete NCT alias)
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-09

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Ablation; Thoracoscopy; Atrial function
MeSH Terms: conditions — Atrial Fibrillation | interventions — Heart Rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endoscopic ablation of atrial fibrillation (Experimental)
  Interventions: Procedure: Endoscopic ablation of AF
- Rate control (Active Comparator)
  Interventions: Drug: Rate control

INTERVENTIONS:
Procedure: Endoscopic ablation of AF — The procedure is conducted in general anaesthesia. The right chest is entered with three working ports .
  After a complete cycle of ablation creating a box lesion in the left atrium, conduction block is tested. A chest tube is placed through the most caudal port and the port incisions are closed. A Reveal loop recorder is then implanted subcutaneously. The patient is extubated and transferred to postoperative care.
  Arms: Endoscopic ablation of atrial fibrillation
Drug: Rate control — Anti-arrhythmic protocol The control group is using a rate-control strategy. All patients keep their anti-arrhythmic/beta-blocker/digoxin medication during the entire follow-up. No attempts are made to rhythm-control the patients, unless subjective symptoms make it necessary.
  Arms: Rate control

SUMMARY:
Primary Objective To evaluate the efficiency of totally endoscopic ablation of AF compared to rate control management of AF.

Secondary Objectives

Does totally endoscopic ablation:

* reduce atrial fibrillation symptoms?
* increase working capacity and improve quality of life?
* improve atrial function?
* reduce the risk for stroke?

DETAILED DESCRIPTION:
This is a randomized open controlled single centre study that involves 60 patients (men and women) over the age of 50 years with longstanding persistent AF of more than one year duration and in the absence of other severe cardiopulmonary disease. One of the participating investigators informs the patient, both verbally and in writing, about the study and what participation in the study involves. The patient will be given time to ask questions and to consider study participation and can be enrolled in the study after signing and dating written Informed Consent. Study duration per patient is 12 months.

After inclusion, the patient will be divided into one of two groups, treatment group or control group, according to block wise randomization. The patient will be asked to complete two health related questionnaires SF 36 and SCL and a transthoracic echocardiography will be conducted together with an exercise test.

The patients will thereafter be assessed according to randomisation. Irrespective of group, the patients will be rescheduled for a visit within two months for totally endoscopic ablation and Reveal implantation or just Reveal implantation (control group). All patients will then be assessed during follow-ups after 1, 3, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 50 years
2. Longstanding persistent AF of > 1 year duration
3. Severe symptoms related to AF
4. Have signed and dated Informed Consent.
5. Willing and able to comply with the protocol for the duration of the trial.

Exclusion Criteria:

1. Severe ischemic heart disease or heart valve disease
2. Thrombus formation in left atrial appendage
3. Intolerance to warfarin medication
4. Advanced pulmonary disease, FEV 1 < 1.5 litre
5. Left atrial diameter > 60 mm
6. Body Mass Index (BMI) > 35 kg/m2
7. Previous pulmonary or heart surgery
8. Participation in another clinical trial within the last 30 days prior to enrollment

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-11; Primary Completion 2014-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Freedom of AF 3 - 12 months postoperatively without antiarrhythmic drugs | 3-12 months

SECONDARY OUTCOMES:
Freedom of symptomatic AF episodes 3 - 12 months | 3-12 months
Exercise capacity after 12 months | 12 months
Quality-of-life assessment (SF-36 and SCL) 3, 6 and 12 months | 12 months
Atrial function and dimensions after 6 and 12 months | 12 months
Freedom of thromboembolic events during the study | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Anders Ahlsson, MD PhD, Principal Investigator — Department of Cardiothoracic Surgery; Espen Fengsrud, MD, Study Chair — Department of Cardiology; Anders Englund, MD PhD, Study Director — Stockholm Arrhythmia Center; Peter Linde, MD, Study Chair — Department of Cardiology; Henrik Almroth, MD, Study Chair — Department of Cardiology; Tommy Andersson, MD, Study Chair — Department of Cardiology; Hans Tyden, MD PhD, Study Chair — Department of Cardiothoracic Surgery
Locations (1):
- Örebro University Hospital, Örebro, Sweden

REFERENCES:
- [Background] Fuster V, Ryden LE, Cannom DS, Crijns HJ, Curtis AB, Ellenbogen KA, Halperin JL, Le Heuzey JY, Kay GN, Lowe JE, Olsson SB, Prystowsky EN, Tamargo JL, Wann S; Task Force on Practice Guidelines, American College of Cardiology/American Heart Association; Committee for Practice Guidelines, European Society of Cardiology; European Heart Rhythm Association; Heart Rhythm Society. ACC/AHA/ESC 2006 guidelines for the management of patients with atrial fibrillation-executive summary: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the European Society of Cardiology Committee for Practice Guidelines (Writing Committee to Revise the 2001 Guidelines for the Management of Patients with Atrial Fibrillation). Eur Heart J. 2006 Aug;27(16):1979-2030. doi: 10.1093/eurheartj/ehl176. No abstract available. PMID 16885201
- [Background] European Heart Rhythm Association (EHRA); European Cardiac Arrhythmia Scoiety (ECAS); American College of Cardiology (ACC); American Heart Association (AHA); Society of Thoracic Surgeons (STS); Calkins H, Brugada J, Packer DL, Cappato R, Chen SA, Crijns HJ, Damiano RJ Jr, Davies DW, Haines DE, Haissaguerre M, Iesaka Y, Jackman W, Jais P, Kottkamp H, Kuck KH, Lindsay BD, Marchlinski FE, McCarthy PM, Mont JL, Morady F, Nademanee K, Natale A, Pappone C, Prystowsky E, Raviele A, Ruskin JN, Shemin RJ. HRS/EHRA/ECAS expert Consensus Statement on catheter and surgical ablation of atrial fibrillation: recommendations for personnel, policy, procedures and follow-up. A report of the Heart Rhythm Society (HRS) Task Force on catheter and surgical ablation of atrial fibrillation. Heart Rhythm. 2007 Jun;4(6):816-61. doi: 10.1016/j.hrthm.2007.04.005. Epub 2007 Apr 30. No abstract available. PMID 17556213
- [Background] Matsutani N, Takase B, Ozeki Y, Maehara T, Lee R. Minimally invasive cardiothoracic surgery for atrial fibrillation: a combined Japan-US experience. Circ J. 2008 Mar;72(3):434-6. doi: 10.1253/circj.72.434. PMID 18296841
- [Background] Sagbas E, Akpinar B, Sanisoglu I, Caynak B, Tamtekin B, Oral K, Onan B. Video-assisted bilateral epicardial pulmonary vein isolation for the treatment of lone atrial fibrillation. Ann Thorac Surg. 2007 May;83(5):1724-30. doi: 10.1016/j.athoracsur.2006.12.009. PMID 17462389
- [Background] Wolf RK, Schneeberger EW, Osterday R, Miller D, Merrill W, Flege JB Jr, Gillinov AM. Video-assisted bilateral pulmonary vein isolation and left atrial appendage exclusion for atrial fibrillation. J Thorac Cardiovasc Surg. 2005 Sep;130(3):797-802. doi: 10.1016/j.jtcvs.2005.03.041. PMID 16153931
- [Background] La Meir M, De Roy L, Blommaert D, Buche M. Treatment of lone atrial fibrillation with a right thoracoscopic approach. Ann Thorac Surg. 2007 Jun;83(6):2244-5. doi: 10.1016/j.athoracsur.2006.08.004. PMID 17532447
- [Derived] Fengsrud E, Wickbom A, Almroth H, Englund A, Ahlsson A. Total endoscopic ablation of patients with long-standing persistent atrial fibrillation: a randomized controlled study. Interact Cardiovasc Thorac Surg. 2016 Aug;23(2):292-8. doi: 10.1093/icvts/ivw088. Epub 2016 Apr 10. PMID 27068249